CLINICAL TRIAL: NCT06159738
Title: The Role of Parental Cognitions in Predicting Wellbeing in Adolescence
Brief Title: Parental Cognitions and Children's Wellbeing
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC21089
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Development
Keywords: wellbeing; parental cognitions; resilience; coping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The current study aims to address the research limitations in previous studies by adopting a longitudinal design to investigate the associations between parental cognitions (parental expectations, parental beliefs, and parental attributional styles) and adolescents' wellbeing, resilience, and coping strategies across an extended period. Two main research questions were posed: 1) What are the associations between parental cognition factors (parental attribution, parental expectations, and parental beliefs and adolescents' outcomes (wellbeing, resilience, and stress-coping)? 2) Which parental cognition factor has the highest probability in predicting the changes of adolescents' wellbeing, resilience, and coping strategies over time? To answer these research questions, bayesian regression analysis was used to identify the best fitting model of adolescents' wellbeing outcomes and to discern the risk and protective roles of parental cognition factors within the model. Bayesian regression approach also enables the assignment of probabilities to each parental cognition factor, quantifying their credibly in relation to adolescents' wellbeing outcomes.

DETAILED DESCRIPTION:
93 parents who has an adolescent aged between 11 to 16 years old were recruited. Only 65 of them had their adolescents to agree to sign up. This result in a 65 dyads of parents and adolescents in total. Parents and adolescents completed the measures on Qualtrics online survey site, respectively. After completion, researcher contacted parents to arrange a zoom call/phone call with their adolescents to complete measures on wellbeing and perceived stress. Among 93 parents who signed up the research, only 65 of their adolescents managed to complete both the online questionnaire and the call with the researcher at baseline. Six months after baseline, only adolescents were asked to repeat the above procedures as the follow-up. 37 adolescents completed the follow-up procedure, which makes this study sample ended up with 37 dyads of parents and adolescents. The primary objective of this observational study is to determine which parental factor, among the three primary parental cognition schemas (parental expectations, parental beliefs, and parental attributional styles), exhibits consistent effects on predicting the changes of adolescents' wellbeing over time.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for participation were parents and their adolescents aged 11 to 16 years old who have no neurodevelopmental conditions reported by parents (specifically to developmental disorders that may include learning difficulties, such as ASD, ADHD, and intellectual disability).

Exclusion Criteria:

* Adolescents with neurodevelopmental disorders, adolescents aged younger than 11 years old or older than 16 years old, and adolescents and parents who are not fluent in English will also be excluded as the measurements in this study are written in English.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 93 parents who has an adolescent aged between 11 to 16 years old were recruited. Only 65 of them had their adolescents to agree to sign up. This result in a 65 dyads of parents and adolescents in total. 39 of them were recruited through secondary state schools, primary state schools, and independent schools in Scotland, England, and Ireland. 15 participants were recruited through a Parent Webinar hosted by the research team. 6 participants were recruited from parenting and child organisations (Glasgow City Parents Group, Shared Parenting Scotland, Connect Scotland, Parental Minds, and the LUNA Project). 5 participants were recruited through research social account on Facebook and Twitter.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Wellbeing | 6 months
  Adolescents' wellbeing (quality of life) measured by KIDCSREEN-27
Resilience | 6 months
  Adolescents' trait resilience measured by Conner Davidson Resilience Scale
Coping Styles | 6 months
  Adolescents' coping styles measured by Brief Coping Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hungtzu Tai, Principal Investigator — University of Edinburgh
Locations (1):
- The University of Edinburgh, Edinburgh, United Kingdom